CLINICAL TRIAL: NCT01661530
Title: A Double Blind Randomised Placebo Controlled Pilot Study of a Dietary Soup Intervention During Pregnancy to Optimise Dietary Vitamin E Intake in Relation to Childhood Asthma.
Brief Title: Piloting a Dietary Vitamin E Intervention During Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2/0036/12; 12/NS/0053 (Other: North of Scotland Research Ethics Service)
Record Dates: First submitted 2012-08-07; First posted 2012-08-09 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Asthma
Keywords: asthma; pregnancy; diet; vitamin E
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin E enhanced diet (Experimental): Range of three vitamin E enhanced soups (400g/tin) containing 18-20mg vitamin in natural food form. Three portions per week
  Interventions: Dietary Supplement: Vitamin E enhanced soup
- Non-enhanced dietary intervention (Placebo Comparator): Range of three similar looking and tasting soups (400g/tin) with naturally low (<3mg) vitamin E content. Three portions per week
  Interventions: Dietary Supplement: Non-enhanced soups

INTERVENTIONS:
Dietary Supplement: Vitamin E enhanced soup — vitamin E enhancement is by virtue of the natural vitamin E content of the food ingredients
  Arms: Vitamin E enhanced diet
Dietary Supplement: Non-enhanced soups — Similar looking and tasting soups with low vitamin E content by virtue of food ingredients
  Arms: Non-enhanced dietary intervention

SUMMARY:
In the last forty years the prevalence of asthma has increased in westernised countries. We have hypothesised that this increase may be a consequence of changing diet. Several birth cohort studies have now reported an association between reduced maternal vitamin E intake during pregnancy and childhood asthma.

However, it remains to be seen whether increasing maternal vitamin E intake during pregnancy reduces the risk of childhood asthma. We are planning a large placebo controlled trial in pregnant women, to investigate whether optimisation of dietary vitamin E intake to the recommended 15mg/day reduces the likelihood of childhood asthma. We believe that a dietary intervention using vitamin E in its natural form of food is more likely to be successful and acceptable than a vitamin E supplement. We have previously demonstrated than pregnant women can optimise their vitamin E intake using a personalised dietary plan with the help of a dietitian however this intervention was complex and could not be translated into everyday use. With commercial support we have developed a range of soups containing foods naturally rich in vitamin E designed to optimise maternal vitamin E intake to 15mg/day. A range of similar tasting and looking placebo soups has also been developed. In this study we will pilot a randomised controlled trial of the active and placebo soups to ascertain whether pregnant women are willing and able to optimise their vitamin E intake during pregnancy using the soups in order to reduce the risk of their child developing asthma. optimising maternal vitamin E intake during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* 10-12 weeks pregnant.
* Routine low risk antenatal care.
* A personal or partner history of asthma at anytime.
* Able and willing to give informed consent to participate
* Able and willing to participate in the study procedures

Exclusion Criteria:

* Use of vitamin E supplements.
* A history of diabetes, coagulopathies or use of anticoagulants, use of clopidogrel, cholestyramine, cyclosporin A, gemfibrozil, isoniazid, orlistat, anticonvulsants.
* Any other significant disease or disorder which, in the opinion of the investigator, either puts the woman at risk because of participating in the study or may influence the results of the study, or the woman's ability to participate in the study.
* Participating in another clinical study
* Previous allocation of randomisation code in the study.

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 59 (Actual)
Dates: Start 2012-12; Primary Completion 2013-06 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Participation of pregnant women in a randomised trial of enhanced and placebo soups from 12 weeks gestation until delivery. | 1 year

SECONDARY OUTCOMES:
Dietary vitamin E intake during pregnancy. | 1 year
Lung function of new born infants. | 1 year

OTHER OUTCOMES:
Biomarker of dietary compliance | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Graham Devereux, MD, Principal Investigator — University of Aberdeen
Locations (1):
- Aberdeen Maternity Hospital, Aberdeen, Aberdeen, United Kingdom

REFERENCES:
- [Background] Devereux G, Turner SW, Craig LC, McNeill G, Martindale S, Harbour PJ, Helms PJ, Seaton A. Low maternal vitamin E intake during pregnancy is associated with asthma in 5-year-old children. Am J Respir Crit Care Med. 2006 Sep 1;174(5):499-507. doi: 10.1164/rccm.200512-1946OC. Epub 2006 Jun 8. PMID 16763215
- [Background] Litonjua AA, Rifas-Shiman SL, Ly NP, Tantisira KG, Rich-Edwards JW, Camargo CA Jr, Weiss ST, Gillman MW, Gold DR. Maternal antioxidant intake in pregnancy and wheezing illnesses in children at 2 y of age. Am J Clin Nutr. 2006 Oct;84(4):903-11. doi: 10.1093/ajcn/84.4.903. PMID 17023719